CLINICAL TRIAL: NCT02212093
Title: Cause-specific 5 Years Mortality-rate in Patients Treated for Severe Pneumonia in an ICU - a Retrospective Study
Brief Title: 5 Years Mortality-rate in Patients Treated for Severe Pneumonia in an ICU - a Retrospective Study
Acronym: pneumonia
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Vegard Dahl, Professor, University Hospital, Akershus
Other Study IDs: 2013/2338
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Pneumonia
Keywords: Pneumonia, mechanical ventilation, ICU, mortality
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Bacteriology tests
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pneumonia and mechanical ventilation: The data are collected retrospectively from this one group.

SUMMARY:
Severe pneumonia has a high in-hospital mortality. There are few studies which investigate the long-term mortality in patients that are discharged alive from the hospital. In this study we want to investigate the 5 years mortality after treatment of severe pneumonia in an ICU. We will also investigate the cause of death after discharge from the hospital.

DETAILED DESCRIPTION:
Patients with severe pneumonia who need treatment in an ICU have a high in-hospital mortality (16-46%). There are few studies which investigate the long-term mortality (> 1year) in patients after discharge from the hospital. There seems to be a higher mortality in this group compared to the general population. The cause(s) of this higher long-term mortality is unclear and few studies have investigated this problem.

We are going to investigate the 5 years mortality rate in this population of patients. We are also going to investigate the cause of death in the patients who are discharged from the hospital alive.

Inclusion criteria: Patients > 18 years. Primary diagnose: pneumonia, and the need of mechanical ventilation for at least 24 hours in an ICU. The patients who arrive at the ICU in Akershus University Hospital in the period from 01.01.1997 to 31.12.2006.

The datas are collected from the patients' journals and the local ICU register. Collecting data: Age, sex, comorbidity, SAPSII, mechanical ventilation time, stay in the ICU, stay in the hospital, ICU mortality, hospital mortality, 5 years mortality, type of pneumonia (bacteriology).

Time of death after discharge is collected from Norwegian National Registry. Cause of death after discharge is collected from Norwegian Institute of Public Health.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years. Primary diagnose: pneumonia, and the need of mechanical ventilation for at least 24 hours in an ICU. The patients who arrived the ICU in Akershus University Hospital in the period from 01.01.1997 to 31.12.2006.

Exclusion Criteria:

* Patients < 18 years. Patients with need for mechanical ventilation < 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The same as the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
5 years mortality | 5 years

SECONDARY OUTCOMES:
cause of death after discharge from the hospital | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Dahl, Professor, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Nordbyhagen, Akershus, Norway